CLINICAL TRIAL: NCT04080037
Title: Assessing Opioid Care Practices Using CPV Patient Simulation Modules to Improve Alignment With CDC Guidelines
Brief Title: Assessing Opioid Care Practices Using CPV Patient Simulation Modules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Ascend Learning (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 01-QALM-2019
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Pain; Pain, Acute; Pain, Chronic; Pain, Neuropathic; Opioid-use Disorder; Opioid Abuse and Addiction; Opioid Withdrawal
MeSH Terms: conditions — Pain; Acute Pain; Chronic Pain; Neuralgia; Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: The study will enroll practicing PCPs in the US. All eligible and consented participants will complete a multiple-choice pre-assessment, the complete 6 weekly patient simulations with feedback and peer benchmarking, then complete a multiple-choice post-assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): All eligible and consented participants will be asked complete a multiple-choice opioid assessment based on the latest CDC opioid guidelines, then care for 6 online QualityIQ patient simulations and receive feedback on their care decisions. They will then all complete an other multiple-choice assessment at the conclusion of the study.
  Interventions: Other: Quality IQ Patient Simulations

INTERVENTIONS:
Other: Quality IQ Patient Simulations — Online patient cases designed to simulate typical patients seen in a primary care practice. In each case, providers will answer multiple-choice questions about their preferred course of action to work-up, diagnose and treat patients in the primary care setting. After each question, providers will receive evidence-based feedback, including references, on the appropriateness of each of their care decisions. Feedback will be supported with relevant reference to evidence-based guidelines, with a specific focus on the CDC opioid guidelines.
  Cases will cover typical primary care patients presenting with acute and chronic pain, who may or may not be already taking opioid medication.
  Other Names: Clinical Performance and Value Vignettes; CPVs

SUMMARY:
This study will test the quality of opioid-related physician care decisions using a patient-simulation based measurement and feedback approach that combines multiple-choice care decisions with real-time, personalized scoring and feedback. The cases and feedback have been designed to align with the latest CDC opioid guidelines. The study will also measure the impact of gaming-inspired competition and motivation, including a weekly leaderboard, to improve evidence-based care decisions. The quality of care decisions will be measured in the simulations and in a multiple-choice assessment administered before and after the patient simulations.

DETAILED DESCRIPTION:
Primary care providers (PCPs) are often on the front lines of helping patients manage acute and chronic pain. These pain management decisions have become especially important in light of the national opioid crisis that has seen an unsettling rise in opioid dependency, over-doses and fatalities. The Centers for Disease Control has developed specific evidence-based guidelines to help clinicians make more informed decisions about appropriate use of opioids as well as identifying and managing patients at risk for opioid-use disorder and overdose.

The investigators' previous work has shown that patient simulations can rapidly and reliably measure unwarranted practice variation among providers. In addition, published work shows that patient simulations, when administered serially and combined with customized feedback on improvement opportunities can reduce practice variation and improve performance on patient-level quality measures. Given the challenge of the current opioid crisis and the large scope of unwarranted variation in medical practice, there is a need for scalable approaches to measure care decisions, provide feedback on improvement opportunities and benchmark performance to peers.

This study seeks to evaluate the impact of personalized measurement and feedback on evidence-based care decisions made by primary care providers across the country concerning opioid care. The study, a prospective cohort trial, will enroll primary care physicians (PCPs) practicing in the U.S. Upon enrollment, eligible providers will be asked to complete a questionnaire detailing their practice and professional background. They will then be asked to complete the following:

Pretest: Pre-project, participants will take a multiple-choice assessment test. These assessments measure CDC Opioid Guidelines knowledge and adherence. Study administrators will randomize half of providers to take Assessment A pre-intervention, and half to take Assessment B pre-intervention, and have attempted to make these two assessments of equal difficulty.

Intervention: All providers will then care for 1 online CPV QualityIQ patient simulation each week over the course of 6 weeks. The simulated patients will be adults aged 18-75 and present with clinical conditions commonly seen by PCPs, such as chronic or acute pain, for whom opioids are currently in use or may be considered. In the patient simulations, participants will make work-up, diagnostic and treatment decisions relevant to the patient's pain management and will receive real-time feedback on how those decisions align with the CDC recommendations. Each week, participants will receive an email notification with their case score from the previous week, how their care compares to their PCP peers, and a link their new case to be completed.

Posttest: Recruits will take the remaining assessment as described above after completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified in internal medicine or family medicine
2. Minimum patient panel size of 1,000 patients
3. At least 5% of their patients currently or previously using opioid medications
4. English-speaking
5. Access to the internet
6. Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

1. Not board certified in either internal medicine or family medicine
2. Patient panel size less than 1,000 patients
3. Less than 5% of their patients currently or previously using opioid medications
4. Non-English speaking
5. Unable to access the internet
6. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Change in provider scores on pre- and post-intervention assessments | 2 months
  At the beginning and end of the study, participants with complete a 20 multiple-choice question assessment to measure familiarity with the latest CDC opioid guidelines. The assessment scales are known as the "QURE-Ascend Learning Modules: Opioids, Assessment A" and "QURE-Ascend Learning Modules: Opioids, Assessment B," both of which measure familiarity with the latest CDC guidelines via multiple-choice questions. Scores on the scales range from 0 to 100%, with a higher score representing greater familiarity with evidence-based care. There are no subscales within the measures.
  Between the assessment, they will care for online simulated patients and receive feedback on their care decisions. A primary outcome in the study will be to measure whether performance on the assessments improves after caring for the simulated patients and receiving feedback. Higher scores on the second assessment represent a better outcome.
Change in the overall and the diagnostic and treatment quality scores in the CPV QualityIQ patient simulations. | 2 months
  In each case, participants will answer multiple-choice questions about their preferred course of action to work-up, diagnose and treat patients in the primary care setting. Each question has specific evidence-based scoring criteria identifying necessary and unnecessary care decisions. Each provider will get a score for each case, ranging from 0 to 100 percentage based on the care decisions they make in the case. Over the course of the project, the investigators will track the percentage of correct, evidence-based care decisions made by participants, with the hypothesis that serial measurement and feedback on evidence-based care decisions will lead to increases in appropriate decisions over time. Higher scores represent a better outcome.

SECONDARY OUTCOMES:
Participant satisfaction as measured by post-evaluation survey | 2 months
  Investigators will measure participant satisfaction as measured by post-evaluation survey. On a scale of 1 to 5 (with 5 being the highest), participants will be asked about the overall quality of the material, the relevance to their practice and the educational content. Higher scores represent a better outcome.
Physician engagement throughout the study | 2 months
  The investigators will track the percentage of enrolled participants who stay engaged in the study and complete at least 80% of their patient simulation cases.

CONTACTS AND LOCATIONS:
Overall Officials: John Peabody, MD, PhD, Principal Investigator — QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers. Analysis will be conducted at the aggregate group level.

REFERENCES:
- [Background] Burgon TB, Cox-Chapman J, Czarnecki C, Kropp R, Guerriere R, Paculdo D, Peabody JW. Engaging Primary Care Providers to Reduce Unwanted Clinical Variation and Support ACO Cost and Quality Goals: A Unique Provider-Payer Collaboration. Popul Health Manag. 2019 Aug;22(4):321-329. doi: 10.1089/pop.2018.0111. Epub 2018 Oct 17. PMID 30328782
- [Background] Weigel PA, Ullrich F, Shane DM, Mueller KJ. Variation in Primary Care Service Patterns by Rural-Urban Location. J Rural Health. 2016 Spring;32(2):196-203. doi: 10.1111/jrh.12146. Epub 2015 Sep 16. PMID 26376210
- [Background] Peabody JW, Luck J, Glassman P, Dresselhaus TR, Lee M. Comparison of vignettes, standardized patients, and chart abstraction: a prospective validation study of 3 methods for measuring quality. JAMA. 2000 Apr 5;283(13):1715-22. doi: 10.1001/jama.283.13.1715. PMID 10755498
- [Background] Peabody JW, Luck J, Glassman P, Jain S, Hansen J, Spell M, Lee M. Measuring the quality of physician practice by using clinical vignettes: a prospective validation study. Ann Intern Med. 2004 Nov 16;141(10):771-80. doi: 10.7326/0003-4819-141-10-200411160-00008. PMID 15545677
- [Background] Schieber LZ, Guy GP Jr, Seth P, Young R, Mattson CL, Mikosz CA, Schieber RA. Trends and Patterns of Geographic Variation in Opioid Prescribing Practices by State, United States, 2006-2017. JAMA Netw Open. 2019 Mar 1;2(3):e190665. doi: 10.1001/jamanetworkopen.2019.0665. PMID 30874783